CLINICAL TRIAL: NCT03696771
Title: A Phase I, Multicenter, Open-label Dose Finding Study of NJH395, Administered Intravenously in Patients With Non-breast HER2+ Advanced Malignancies
Brief Title: Study to Determine Safety and Dose of NJH395 in Non-breast HER2+ Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNJH395X2101
Record Dates: First submitted 2018-09-04; First posted 2018-10-05 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: NON-breast HER2+ Malignancies
Keywords: Phase I, NJH395, HER2+, ISAC, TLR7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NJH395 (Experimental): Includes non-breast HER2-positive advanced malignancies
  Interventions: Drug: NJH395

INTERVENTIONS:
Drug: NJH395 — Immune stimulator antibody conjugate (ISAC), consisting of a monoclonal antibody which targets HER2 conjugated to an immune-stimulatory agent

SUMMARY:
A first-in-human study using NJH395 in non-breast HER2-positive advanced malignancies

DETAILED DESCRIPTION:
This study has two parts. There will be a single dose of NJH395 in the first part and multiple doses of NJH395 in the second part. After the first part is completed, the second part may open.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient must have known histologically or cytologically confirmed and documented HER2-positive solid tumor excluding patients with breast cancer
* Advanced/metastatic cancer with measurable disease as determined by RECIST v.1.1 who have progressed or are intolerant to all approved therapies known to confer clinical benefit.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Patient must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Patient must be willing to undergo a new tumor biopsy prior to therapy, and during therapy on this study.

Key Exclusion Criteria:

* History of severe hypersensitivity to any ingredient of study drug, trastuzumab or other monoclonal antibody.
* Patients previously treated with TLR 7/8 agonist.
* Impaired cardiac function or history of clinically significant cardiac disease
* Active, known or suspected autoimmune disease.
* Human Immunodeficiency virus (HIV) infection
* History of or current interstitial lung disease or pneumonitis Grade 2 or greater.
* Discontinued prior checkpoint inhibitor due to a checkpoint inhibitor related toxicity.
* Currently receiving medications known to cause Torsades de Pointe that cannot be discontinued 7 days prior to starting treatment

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities (DLTs) | 21 days
  The time frame will expand to 42 days for the second part of the study
Number of participants with Adverse Events | 2.5 years

SECONDARY OUTCOMES:
Concentration versus time profiles for NJH395 and its catabolite | 126 days
PK parameter (Cmax) for NJH395 | 126 days
Pharmacokinetic (PK) parameter (AUC) for NJH395 | 126 days
Incidence of anti-NJH395 antibodies and neutralizing antibodies to trastuzumab | 126 days
Overall Response Rate | 2.5 years
  Response assessed by RECIST v1.1 and iRECIST
Clinical Benefit Rate (CBR) | 2.5 years
  Response assessed by RECIST v1.1 and iRECIST
Progression Free Survival (PFS) | 2.5 years
  Time from start of treatment to date of the first documented progression or death in months
Duration of Response (DOR) | 2.5 years
  Response assessed by RECIST v1.1 and iRECIST
Characterization of tumor-infiltrating lymphocytes by IHC | Cycle 1 Day 5, Cycle 2 Day 1 (each cycle is 21 days), Cycle 8 Day 1 and at end of treatment (expected between months 6 and 7)
  Change from baseline in TILs by immunohistochemistry (IHC) (such as CD8).

CONTACTS AND LOCATIONS:
Locations (4):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Novartis Investigative Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janku F, Han SW, Doi T, Amatu A, Ajani JA, Kuboki Y, Cortez A, Cellitti SE, Mahling PC, Subramanian K, Schoenfeld HA, Choi SM, Iaconis LA, Lee LH, Pelletier MR, Dranoff G, Askoxylakis V, Siena S. Preclinical Characterization and Phase I Study of an Anti-HER2-TLR7 Immune-Stimulator Antibody Conjugate in Patients with HER2+ Malignancies. Cancer Immunol Res. 2022 Dec 2;10(12):1441-1461. doi: 10.1158/2326-6066.CIR-21-0722. PMID 36129967
- See also: Plain language summaries are available on this link — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=970